CLINICAL TRIAL: NCT04660591
Title: Cemented Long Versus Standard Femoral Stem Arthroplasty for Proximal Femoral Metastasis
Brief Title: Length of the Femoral Stem in Arthroplasty Done for Patients With Proximal Femoral Metastatic Lesion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ibrahim Mahmoud Abdelmonem, Dr, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU MD 277/ 2019
Record Dates: First submitted 2020-11-27; First posted 2020-12-09 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Metastatic Bone Tumor; Pathological Fracture; Arthroplasty
Keywords: pathological, metastasis ,; cement reaction; long stem
MeSH Terms: conditions — Bone Neoplasms; Fractures, Spontaneous; Neoplasm Metastasis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Intervention Model Description: two comparative groups, standard and long femoral stem arthroplasty
Who Masked: Participant
Masking Description: only participants were blinded from treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- standard femoral stem (Active Comparator): standard length femoral stem arthroplasty applied for patients with proximal femoral metastasis either impending or pathological fracture
  Interventions: Device: femoral stem in hip arthroplasty
- long femoral stem (Active Comparator): long femoral stem arthroplasty applied for patients with proximal femoral metastasis either impending or pathological fracture
  Interventions: Device: femoral stem in hip arthroplasty

INTERVENTIONS:
Device: femoral stem in hip arthroplasty — using lateral approach to the hip we will compare the effect of femoral stem length on the oncological and functional outcomes in patients with proximal femoral metastasis.hip arthroplasty is a surgical procedure that involves changing the head of the femur (the ball) with or without replacing the articular surface of the acetabulum (the socket ).and replacing it with metal head based on a stem covered with cement to fix it to the bone of the femur.
  Other Names: cemented hip arthroplasty , hip replacement

SUMMARY:
Proximal femoral metastatic disease is a common cause of morbidity and mortality in cancer patients.protecting the entire femur using long nail or long femoral stem was hypothesized to prevent future fracture.However we believe that long stem isn't always necessary and won't decrease the complication rate.noting it's increased complication rate in this high risk patient category .

DETAILED DESCRIPTION:
Skeletal metastasis is the third most common site of cancer metastasis after the lungs and liver, almost all patients with metastatic prostate cancer will have bone metastasis. And about 90% of patients dying from breast cancer has skeletal metastasis.

The most common site to which cancer metastasize to long bones is the proximal femur, especially to the intertrochanteric region and femoral neck, contributing to increasing incidence of impending and pathologic fractures of this site.(8) Recent advances in cancer treatment increased the longevity of patients, with subsequent increase in morbidity of metastatic disease and increased number of patients living longer with this condition .

To date, long femoral stem is most frequently used in cases of pathological and impending proximal femoral fractures. Its use is believed to add more stability and prophylactically protect the entire femur from newly developed distal lesions. However, long stems has more operative time, more cardiopulmonary complications and are more technically demanding compared to standard femoral stems arthroplasty.(5) Recent retrospective study by Xing et al reported comparable outcomes between standard, medium and long stems and concluded that the routine use of long stems is unjustified.Another recent report by Joel et al investigated the use of long femoral stem in 22 limbs, they reported no hardware failure with no cases of intraoperative cardiopulmonary complications, however they recommended larger comparative trials with rigorous methods to investigate the functional outcomes and complications of long femoral stems in proximal femoral metastatic lesions.

In face of the potential advantages in this patient population, the goal of this study is to investigate the use of standard length femoral stems and its results compared to long femoral stems in proximal femoral metastasis .

ELIGIBILITY:
Inclusion Criteria:

* pathological or impending pathological pertrochanteric or neck femur fracture, regardless of the presence of distal femoral metastasis.

Exclusion Criteria:

* Previous arthroplasty in the same side. fractures or lesions involving the subtrochanteric region Pathological fracture due to metabolic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
MSTS score | Implant-specific differences in postoperative functional outcomes will be determined and compared throughout the study period at different time points(preoperative, postoperative at one month, six months and one year)
  The Musculoskeletal Tumor Society (MSTS) scoring system is a disease-specific instrument to determine the physical and mental health for patients with extremity sarcoma
survival | Implant-specific differences in survival will be determined and compared throughout the study period at different time points(preoperative, postoperative at one month, six months and one year)
  median and mean patient survival

SECONDARY OUTCOMES:
visual analogue score | improvement of pain compared to preoperative status
  VAS as a measure for pain relief
the Eastern Cooperative Oncology Group (ECOG) Scale of Performance Status | implant specific ECOG as a measure of patient functional level compared at different time points(preoperative ,one month ,six months and one year postoperative)
  is a simple measure of functional status. It has scores ranging from 0 to 5
complications | will be reported during one year follow up
  postoperative infection (superficial or deep),dislocation

CONTACTS AND LOCATIONS:
Locations (1):
- AinShams university, Cairo, Abbasid, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: after publishing the study no limit regarding how long data will be shared

REFERENCES:
- [Background] Coleman RE. Clinical features of metastatic bone disease and risk of skeletal morbidity. Clin Cancer Res. 2006 Oct 15;12(20 Pt 2):6243s-6249s. doi: 10.1158/1078-0432.CCR-06-0931. PMID 17062708
- [Background] Schneiderbauer MM, von Knoch M, Schleck CD, Harmsen WS, Sim FH, Scully SP. Patient survival after hip arthroplasty for metastatic disease of the hip. J Bone Joint Surg Am. 2004 Aug;86(8):1684-9. doi: 10.2106/00004623-200408000-00011. PMID 15292415
- [Background] Tsuda Y, Yasunaga H, Horiguchi H, Fushimi K, Kawano H, Tanaka S. Complications and Postoperative Mortality Rate After Surgery for Pathological Femur Fracture Related to Bone Metastasis: Analysis of a Nationwide Database. Ann Surg Oncol. 2016 Mar;23(3):801-10. doi: 10.1245/s10434-015-4881-9. Epub 2015 Oct 5. PMID 26438441
- [Background] Xing Z, Moon BS, Satcher RL, Lin PP, Lewis VO. A long femoral stem is not always required in hip arthroplasty for patients with proximal femur metastases. Clin Orthop Relat Res. 2013 May;471(5):1622-7. doi: 10.1007/s11999-013-2790-4. Epub 2013 Jan 30. PMID 23361930
- [Result] Peterson JR, Decilveo AP, O'Connor IT, Golub I, Wittig JC. What Are the Functional Results and Complications With Long Stem Hemiarthroplasty in Patients With Metastases to the Proximal Femur? Clin Orthop Relat Res. 2017 Mar;475(3):745-756. doi: 10.1007/s11999-016-4810-7. PMID 27052019
- [Derived] Abdelmonem IM, Azmy SI, El Masry AM, El Ghazawy AK, Kotb AS, Bassiony AA. Cemented long versus standard femoral stem in proximal femoral metastasis: a noninferiority single-blinded quasi-randomized clinical trial. Eur J Trauma Emerg Surg. 2022 Aug;48(4):2977-2985. doi: 10.1007/s00068-021-01875-x. Epub 2022 Feb 13. PMID 35152311